CLINICAL TRIAL: NCT02987790
Title: Duration of Antibiotic Therapy in Critically Ill Patients: C-reactive Protein-guided Therapy Versus Best Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: Fundação de Amparo à Pesquisa do estado de Minas Gerais (Other)
Responsible Party: Principal Investigator, Vandack Alencar Nobre, PhD, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCRxBestPractice
Record Dates: First submitted 2016-12-05; First posted 2016-12-09 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Infection Systemic
Keywords: Intensive care; Sepsis; Biomarkers; C-reactive Protein; Antimicrobial; Systemic infection
MeSH Terms: conditions — Toxemia; Sepsis | interventions — C-Reactive Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- C-reactive Protein (Experimental): In this group, the attending physicians will be instructed to follow the decision flowchart based on the CRP values. Antibiotic suspension will be encouraged when levels of this marker are <35mg/L (if peak PCR below 100mg/L); or reduce 50% of the highest value (if PCR peak > 100mg/L), with a limit of seven days, if there is clinical improvement. If a given patient has persistently elevated CRP levels (> 100 mg/l or fall less than 50% relative to the time of inclusion), the investigators will encourage attending physicians to maintain antibiotics and to perform a careful search for persistent infection. In case of doubts, if the patient is well clinically and without signs of active infection, the duration of antibiotic therapy should be the same as suggested for the Best Practice group.
  Interventions: Other: C-reactive protein
- Best Practice (No Intervention): Patients will be initially treated according to the current protocols used in the intensive care units. Decisions about interruption or continuation of treatment will be made according to pre-established time and also according to the clinical evolution of the patients. CRP levels will not be measured and will not be considered in the decision to discontinue antimicrobials. Any decision ultimately rests with the clinical assistants. Suggestions on the suspension of antibiotics will be provided by the researchers as follows:
  * 7 full days for most infections
  * 10 full days for pneumonia caused by Gram negative non-fermenting bacteria or Gram negative bacteria carbapenemase producing.
  * 14 days of treatment for necrotizing pneumonia, confirmed by chest computed tomography.

INTERVENTIONS:
Other: C-reactive protein — PCR assays shall be performed daily on serum obtained from blood collected for routine intensive care examinations up to 2 days after antibiotic withdrawal. In the PCR group, antibiotic suspension will be encouraged when levels of this marker are <35mg / L (if peak PCR below 100mg / L); or reduce 50% of the highest value (if PCR peak> 100mg / L), with a limit of seven days, if there is clinical improvement.
  Arms: C-reactive Protein

SUMMARY:
The judicious use of antibiotics is one of the main measures to limit the emergence of multidrug-resistant pathogen related to excessive antimicrobial use. A recent study demonstrated that C-reactive protein (CRP) was as useful as procalcitonin (PCT) in reducing the time of antibiotic therapy in adult septic patients treated in the ICU setting. Therefore, the present study proposes to compare the time of use of antimicrobials, costs of hospitalization and clinical outcomes of interest among a group of antibiotic therapy guided by serum levels of CRP and a group of therapy based on the best practices of antibiotic therapy (Best Practice).

DETAILED DESCRIPTION:
All adult patients (aged> 17 years), hospitalized at the ICU (total of 50 beds) of the Hospital das Clínicas - UFMG, with an assumed or proven infection, will be considered for inclusion. Patients who meet the inclusion and exclusion criteria will be allocated randomly into one of the following groups: 1) PCR group: antibiotic therapy will be discontinued according to serum CRP levels; 2) "Best Practice" group, length of antibiotic therapy based on the most recent guidelines in the medical literature, according to the focus and / or causative micro-organism. PCR assays shall be performed daily on serum obtained from blood collected for routine intensive care examinations up to 2 days after antibiotic withdrawal. In the PCR group, antibiotic suspension will be encouraged when levels of this marker are <35mg / L (if peak PCR below 100mg / L); or reduce 50% of the highest value (if PCR peak > 100mg / L), with a limit of seven days, if there is clinical improvement. Primary outcomes will be duration of antibiotic therapy and antibiotic-free live days corrected for 1000 days of hospitalization. Secondary outcomes will be costs, clinical cure rate, therapeutic failure, 28-day mortality, 90-day mortality, in-hospital mortality, length of hospital stay, nosocomial infection rate, recurrence of infection, and isolation of multidrug-resistant bacteria

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Signed informed consent
* Assumed or proven infection
* Patient admitted to the unit participating in the study

Exclusion Criteria:

* Patients with severe immunosuppression, such as severe neutropenia (<500 neut/mm3), transplantation of solid organs or cells hematopoietic, HIV infection with CD4+ < 200/mm3
* Patients with multiple trauma, burns or surgery grid size in the last 5 days (Except surgery for focus control)
* Use of antibiotics supposedly or proven to be effective against the infectious process in for more than 48 hours.
* Patients undergoing palliative care.
* Patients with death expectancy for the next 24 hours.
* Patients with bacteremia caused by Staphylococcus aureus or Candida spp
* Patients with infections that are known to require prolonged antibiotic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Duration of antibiotic therapy for the first episode of infection | 1 year
  Days of treatment with antibiotics after inclusion
Total antibiotic exposure days per 1,000 days | 1 year

SECONDARY OUTCOMES:
Costs of hospitalization | Through study completion, an average of 1 year
  Considering Brazilian market prices
Clinical cure rate | 28 days
  Disappearance of clinical signs and symptoms present at inclusion
Therapeutic failure | 28 days
  Persistence or recurrence of the pathogen originally causing the infection.
All cause 28-day mortality | 28 days
All cause 90-day mortality | 90 days
Length of ICU stay | 28 days
Length of hospital stay | 28 days
Nosocomial infection rate | 28 days
Isolation of multiresistant bacteria | 28 days
In-hospital mortality | An average of 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Vandack Nobre, PhD, Study Director — Medical School of the Federal University of Minas Gerais; Isabela Borges, MSc, Principal Investigator — Medical School of the Federal University of Minas Gerais
Locations (1):
- Hospital das Clínicas - Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Borges I, Carneiro R, Bergo R, Martins L, Colosimo E, Oliveira C, Saturnino S, Andrade MV, Ravetti C, Nobre V; NIIMI - Nucleo Interdisciplinar de Investigacao em Medicina Intensiva. Duration of antibiotic therapy in critically ill patients: a randomized controlled trial of a clinical and C-reactive protein-based protocol versus an evidence-based best practice strategy without biomarkers. Crit Care. 2020 Jun 1;24(1):281. doi: 10.1186/s13054-020-02946-y. PMID 32487263